CLINICAL TRIAL: NCT06494358
Title: Liquid Biopsies for the Detection of Somatic Mutations in Brain Arteriovenous Malformations
Brief Title: Liquid Biopsies for the Detection of Somatic Mutations in bAVMs
Acronym: BioMAV
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240718
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-04

CONDITIONS: Brain Arterial Disease
Keywords: brain arteriovenous malformation; liquid biopsies
MeSH Terms: conditions — Intracranial Arterial Diseases | interventions — Liquid Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Circulating DNA: There will be 1 tube of 2 mL (arterial sample near the nidus, collected as part of standard care but conserved for research) and 2 tubes of 10 mL (peripheral blood sampled from the care catheter), in addition to the samples taken as part of standard care during the embolization procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: liquid biopsies and surgery specimen analysis — liquid biopsies and surgery specimen analysis

SUMMARY:
"Personalized medicine has revolutionized patient care, particularly in oncology. Brain arteriovenous malformations (bAVMs) are abnormal vessels located on the surface of the brain or within the brain parenchyma, causing abnormal communication between arterial and venous networks, without the interposition of the capillary bed. The main risk of these malformations is rupture, leading to intracranial bleeding, which can cause severe sequelae or even death. bAVMs (except those of clearly identified genetic origin [< 5%], such as mutations associated with Rendu-Osler disease) have long been considered non-genetic in origin.

However, somatic genetic mutations activating the RAS/RAF/MEK/ERK (MAPK) signaling pathway have recently been identified in surgical specimens of bAVMs. Additionally, targeted inhibition of this pathway is effective in treating these malformations in animals and appears to be effective in extracranial arteriovenous malformations, particularly superficial ones.

Next-generation sequencing of circulating DNA on liquid biopsies is a promising and minimally invasive approach to studying the presence of mutations in arteriovenous malformations.

The treatment of a bAVM aims to obliterate the malformation to prevent or avoid the risk of hemorrhage. It may involve several therapeutic modalities: microsurgery, endovascular embolization, and radiosurgery. These treatments can be combined, and microsurgery is often preceded by pre-surgical embolization, aimed at reducing the hemorrhagic risk of the intervention. However, these are invasive treatments, not without risk.

The identification of mutations through liquid biopsies could enable the development of non-invasive targeted therapies against these bAVMs.

This research aims to identify somatic genetic mutations activating the MAPK signaling pathway in bAVMs. These mutations have already been identified in surgical specimens. This research aims to evaluate the diagnostic performances of liquid biopsies (detection of genetic mutations in blood samples, i.e., circulating DNA), with the gold standard being the detection of the same mutations in surgical specimens."

DETAILED DESCRIPTION:
"Description of Domain Knowledge Personalized medicine has revolutionized patient care, especially in oncology. Brain arteriovenous malformations (bAVMs) are abnormal vessels located on the brain's surface or within the cerebral parenchyma, abnormally connecting the arterial and venous networks without the intermediary of the capillary bed. The primary risk of these malformations is rupture, leading to intracranial bleeding, which can cause severe sequelae or even death. bAVMs (excluding those of clearly identified genetic origin [< 5%], such as mutations associated with Rendu-Osler disease) have long been considered non-genetic in origin.

However, somatic genetic mutations activating the RAS/RAF/MEK/ERK (MAPK) signaling pathway have recently been identified in surgical specimens of bAVMs [1]. Moreover, targeted inhibition of this pathway is effective in treating these malformations in animal models [2] and seems effective in extracranial arteriovenous malformations, particularly superficial ones [3].

Next-generation sequencing of circulating DNA on liquid biopsies is a promising new approach, allowing for a non-invasive study of mutations in arteriovenous malformations [4].

The treatment of a bAVM aims to obliterate the malformation to prevent or mitigate hemorrhagic risk. Several therapeutic modalities can be used: microsurgery, endovascular embolization, and radiosurgery. These treatments can be combined, with microsurgery often preceded by pre-surgical embolization to reduce the hemorrhagic risk of the intervention. However, these treatments are invasive and not without risk [5].

The identification of mutations through liquid biopsies would enable the development of non-invasive targeted therapies against these bAVMs [6].

Description of the Population to be Studied and Justification for Their Choice The population consists of patients aged 18 years or older with a bAVM, for whom treatment by microsurgery with preoperative embolization at Pitié-Salpêtrière Hospital was decided upon in a multidisciplinary consultation meeting.

The choice of this particular population (patients treated with embolization followed by surgery) is justified by the need to obtain the gold standard diagnosis on a surgical specimen for the primary evaluation criteria of the study.

Some patients, whose initial decision in the multidisciplinary consultation was treatment by microsurgery with preoperative embolization, will undergo complete embolization. These patients will not have surgery, and the initially planned surgery will be canceled subsequently. These patients will only be included in the analysis of certain secondary outcome criteria. This accounts for about half of the patients.

In total, there will be 25 patients for the primary evaluation criteria and about twice as many for the secondary evaluation criteria.

Description of Research Elements The research focuses on identifying somatic genetic mutations activating the RAS/RAF/MEK/ERK (MAPK) signaling pathway in brain arteriovenous malformations. These mutations have already been identified in surgical specimens. This research aims to evaluate the diagnostic performance of liquid biopsies (search for genetic mutations on blood samples, i.e., circulating DNA search), with the gold standard being the search for the same mutations on surgical specimens.

These liquid biopsies will be performed during the embolization procedure by arterial sampling near the malformation and on peripheral venous blood (no additional procedure compared to usual care). A blood sample taken from the artery immediately adjacent to the nidus (2 mL) will use the aspirated blood to check the microcatheter's patency, according to standard care procedures (normally not conserved sample), and two other blood samples will be taken from a peripheral vein [one at the beginning of the embolization procedure (10 mL) and one at the end of the embolization procedure (10 mL)] via the venous catheter used by the anesthesia team as part of standard care. This tube taken at the end of the procedure is justified by the hypothesis of the release of mutated cells linked to embolization.

Thus, for the research, there will be 1 tube of 2 mL (arterial sample near the nidus, collected as part of standard care but conserved for research) and 2 tubes of 10 mL (peripheral blood sampled from the care catheter), in addition to the samples taken as part of standard care during the embolization procedure.

Primary Objective To study the diagnostic performance of 1) liquid biopsies on the artery near the nidus and 2) liquid biopsies on peripheral veins for identifying somatic genetic mutations in bAVMs compared to the gold standard diagnosis on a surgical specimen.

Secondary Objectives

* Evaluate the prevalence of genetic mutations identified on surgical specimens.
* Evaluate the prevalence of genetic mutations identified by liquid biopsies on the artery near the nidus.
* Evaluate the prevalence of genetic mutations identified by liquid biopsies on peripheral veins.
* Evaluate the general characteristics of patients (age, gender, mode of presentation) for each identified mutation.
* Evaluate imaging characteristics of bAVMs for each identified mutation. Number of Participating Centers Monocentric study
* Recruiting center: Interventional Neuroradiology Unit, Pitié-Salpêtrière Hospital"

ELIGIBILITY:
"_Age ≥ 18 years

* Treated for bAVM at Pitié-Salpêtrière Hospital
* Indication for treatment by embolization followed by surgery decided in a multidisciplinary consultation meeting (RCP) at Pitié-Salpêtrière Hospital
* Treatment by embolization possibly followed by surgery within 24-48 hours if the embolization is incomplete
* Informed about the study and not objecting to participation"

Exclusion criteria :

* Extra-cerebral arteriovenous malformations
* Under legal protection (guardianship/curators, etc.)
* Pregnancy
* Not eligible for combined treatment (embolization followed by surgery)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The population consists of patients aged 18 years or older with a bAVM, for whom treatment by microsurgery with preoperative embolization at Pitié-Salpêtrière Hospital was decided upon in a multidisciplinary consultation meeting.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Study of the diagnostic performance of 1) liquid biopsies on the artery in the immediate vicinity of the nidus, 2) liquid biopsies on the peripheral vein, for the detection of somatic genetic mutations in cAVMs | 18 months
  - Sensitivity / Specificity / Positive Predictive Value / Negative Predictive Value Compared with the gold standard: detection of mutations on surgical specimens

SECONDARY OUTCOMES:
- Prevalence of mutations on surgical specimens | 18 months
- Prevalence of mutations on the artery in the immediate vicinity of the nidus | 18 months
- Prevalence of peripheral vein mutations | 18 months
- General patient characteristics for each of the mutations identified | 18 months
- Imaging characteristics of cAVMs for each of the mutations identified | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Unité de neuroradiologie interventionnelle, hôpital Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients. Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.